CLINICAL TRIAL: NCT03272061
Title: The Effects of Aerobic-based Exercise on Brain Vascular Function in Elderly Men
Brief Title: Exercise and Brain Vascular Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: METC173025
Record Dates: First submitted 2017-08-29; First posted 2017-09-05 (Actual); Last update posted 2019-01-16 (Actual); Status verified 2019-01

CONDITIONS: Physical Exercise; Cerebrovascular Function; Cerebral Blood Flow; Glucose Metabolism; Cognitive Performance
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants will follow in randomized order a tightly controlled, progressive, aerobic-based exercise program or control program for eight weeks, separated by a washout period of twelve weeks.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic-based exercise program (Experimental)
  Interventions: Other: Aerobic-based exercise program
- Control program (No Intervention): Maintenance of habitual physical activity levels

INTERVENTIONS:
Other: Aerobic-based exercise program — Aerobic-based exercise will be carried out on a cycling ergometer three times a week for 30 minutes at 70% of the maximal workload. Every two weeks, the maximal workload will be reassessed, and training loads will be readjusted accordingly. Fully supervised training sessions will be performed with three-to-four study participants at a time. Subjects should maintain their body weight during the intervention period.
  Arms: Aerobic-based exercise program

SUMMARY:
Cognitive performance is negatively related to an impaired glucose metabolism, possibly due to impairments in brain vascular function. Supported by the statement from the American Heart and Stroke Association that physical exercise is one of the most effective strategies to protect against cognitive decline, we now hypothesize that exercise-induced changes in glucose metabolism cause beneficial effects on brain vascular function thereby improving cognitive performance. The primary objective of this intervention study is thus to evaluate in sedentary elderly men the effect of a 8-week aerobic-based exercise program on cerebral blood flow, as quantified by the non-invasive gold standard magnetic resonance imaging (MRI) perfusion method Arterial Spin Labeling (ASL). Cerebral blood flow is a robust and sensitive physiological marker of brain vascular function. Secondary objectives are to examine effects on glucose metabolism using the oral glucose tolerance test and cognitive performance as assessed with a neurophysiological test battery.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 60-70 years
* Men
* BMI between 25-35 kg/m2 (overweight and slightly obese)
* Sedentary (not moderately active for 3 times or more per week)
* Fasting plasma glucose < 7.0 mmol/L
* Fasting serum total cholesterol < 8.0 mmol/L
* Fasting serum triacylglycerol < 4.5 mmol/L
* Systolic blood pressure < 160 mmHg and diastolic blood pressure < 100 mmHg
* Stable body weight (weight gain or loss < 3 kg in the past three months)
* Willingness to give up being a blood donor from 8 weeks before the start of the study, during the study and for 4 weeks after completion of the study
* No difficult venipuncture as evidenced during the screening visit

Exclusion Criteria:

* Women
* Current smoker, or smoking cessation < 12 months
* Diabetic patients
* Familial hypercholesterolemia
* Abuse of drugs
* More than 3 alcoholic consumptions per day
* Use of dietary supplements known to interfere with the main study outcomes as judged by the principal investigators
* Use medication to treat blood pressure, lipid or glucose metabolism
* Use of an investigational product within another biomedical intervention trial within the previous 1-month
* Severe medical conditions that might interfere with the study, such as epilepsy, asthma, kidney failure or renal insufficiency, chronic obstructive pulmonary disease, inflammatory bowel diseases, auto inflammatory diseases and rheumatoid arthritis
* Active cardiovascular disease like congestive heart failure or cardiovascular event, such as an acute myocardial infarction or cerebrovascular accident
* Contra-indications for MRI imaging (e.g. pacemaker, surgical clips/material in body, metal splinter in eye, claustrophobia)

Ages: 60 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Brain vascular function | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  Cerebral blood flow as quantified non-invasively by the MRI perfusion method Arterial Spin Labeling (ASL)

SECONDARY OUTCOMES:
Glucose metabolism | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  Oral Glucose Tolerance Test (OGTT)
Cognitive performance | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  Cambridge Neuropsychological Test Automated Battery (CANTAB)

OTHER OUTCOMES:
Other physiological parameters: Peripheral vascular function | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  Flow-mediated vasodilation (FMD), carotid artery reactivity, pulse wave analysis (PWA) and velocity (PWV), and retinal images
Other physiological parameters: Blood pressure | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  Office and 24-hour ambulatory blood pressure
Other physiological parameters: Continuous blood glucose | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  36-hour glycaemic response
Other physiological parameters: Advanced glycation endproducts | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  Serum protein-bound advanced glycation endproducts (AGEs)
Other physiological parameters: Conventional metabolic risk markers | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  Lipids and lipoproteins, glucose and insulin, and markers for low-grade systemic inflammation and microvascular function
Other perceivable benefits: Quality of Life | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  The Quality of life (QoL) will be assessed using a 32-item questionnaire
Other perceivable benefits: Sleep characteristics | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  Sleep characteristics will be assessed using the 10-item Pittsburgh Sleep Quality Index
Other perceivable benefits: Mood | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  Mood will be tested using the Affect Grid
Other perceivable benefits: Physical fitness (1) | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  Incremental exhaustive exercise test (VO2 max)
Other perceivable benefits: Physical fitness (2) | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  Timed up-and-go test (TUGT)
Other perceivable benefits: Physical fitness (3) | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  The 6-minute walk test (6 MWT)
Other perceivable benefits: Physical fitness (4) | Difference between outcomes at the end of an 8-week aerobic-based exercise and control program
  Handgrip and muscle strength tests

CONTACTS AND LOCATIONS:
Overall Officials: Peter J Joris, PhD, Principal Investigator — Maastricht University Medical Center; Ronald P Mensink, PhD, Principal Investigator — Maastricht University Medical Center
Locations (1):
- Maastricht University Medical Center, Maastricht, Netherlands

REFERENCES:
- [Derived] Mashnafi S, Plat J, Mensink RP, Joris PJ, Kleinloog JPD, Baumgartner S. Effects of an 8-week aerobic exercise program on plasma markers for cholesterol absorption and synthesis in older overweight and obese men. Lipids Health Dis. 2021 Sep 21;20(1):112. doi: 10.1186/s12944-021-01537-2. PMID 34548089
- [Derived] Kleinloog JPD, Mensink RP, Ivanov D, Adam JJ, Uludag K, Joris PJ. Aerobic Exercise Training Improves Cerebral Blood Flow and Executive Function: A Randomized, Controlled Cross-Over Trial in Sedentary Older Men. Front Aging Neurosci. 2019 Dec 4;11:333. doi: 10.3389/fnagi.2019.00333. eCollection 2019. PMID 31866855